CLINICAL TRIAL: NCT03691311
Title: An Open Label Biomarker Pilot Study of the Antitumoral Activity of Denosumab in the Pre- Operative Setting of Early Breast Cancer
Brief Title: Biomarker Study of the Antitumoral Activity of Denosumab in the Pre- Operative Setting of Early Breast Cancer
Acronym: D-BIOMARK
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICO 13-001; 2016-002678-11 (EudraCT Number); 20119112 (Other Grant/Funding Number: Amgen reference)
Record Dates: First submitted 2018-09-04; First posted 2018-10-01 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Breast Neoplasm Female; Stage I Breast Cancer; Stage II Breast Cancer; Hormone Receptor Negative Neoplasm; Hormone Receptor Positive Tumor
Keywords: rank; rankl; denosumab
MeSH Terms: conditions — Breast Neoplasms; Osteopetrosis, Autosomal Recessive 7; Osteopetrosis, mild autosomal recessive form | interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: This is a parallel two arms trial randomized in 2:1 proportions to intervention group vs control group. . At least 24 patients with hormone receptor negative breast cancer and 24 premenopausal patients will be included in the study so allocation of patients without any of these two characteristics will be restricted depending on the overall characteristics of the included population
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab (Experimental): Denosumab 120 MG/1.7 ML Subcutaneous Solution [XGEVA]
  Interventions: Drug: Denosumab 120 MG/1.7 ML Subcutaneous Solution [XGEVA]
- Control (No Intervention): Control group

INTERVENTIONS:
Drug: Denosumab 120 MG/1.7 ML Subcutaneous Solution [XGEVA] — Two injections on days 1 and 8 previous to surgery breast cancer excision
  Arms: Denosumab

SUMMARY:
This is a biomarker study designed to test the preclinically generated hypothesis of anti-tumoral activity of denosumab in patients with early breast cancer candidates a tumour excision

DETAILED DESCRIPTION:
This is a biomarker study designed to test in patients the preclinically generated hypothesis of anti-tumoral activity of denosumab.The main objective is to demonstrate the antiproliferative and/or pro-apoptotic activity of denosumab in early breast cancer. Other endpoints are to correlate denosumab activity with RANK and RANKL expressions through mRNA and protein; to characterize the differential antiproliferative activity of denosumab between different phenotypes of breast cancer; to identify biomarkers, to identify global changes in gene expression and validate the activity of RANKL antibody in clinical samples. A total of 60 patients with early breast cancer (Stages I and II) candidates to tumor excision as first therapeutic approach will be randomized 2:1, a treatment arm that will receive two doses of denosumab following diagnosis, and a control arm that will not receive treatment. At least 24 patients with hormone receptor negative breast cancer and 24 premenopausal patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign Informed Consent for this study.
* Women ≥ than 18 years, (the inclusion process will be modified to recruit at least 24 premenopausal patients).
* Capable, under investigator judgment, to understand the non-therapeutic nature of the study.
* Diagnosed with invasive breast cancer in early, curable, stage (I or II) candidate to radical surgery as first therapeutic approach.
* Her2 negative receptor status.
* Any estrogen, progesterone status (the inclusion process will be modified to recruit at least 24 patients with TNBC tumors).
* No previous systemic treatment for any malignancy.
* No ongoing treatment with denosumab or bisphosphonates.
* Tumour amenable for baseline Biopsy and punch-Biopsy after excision.

  * Adequate Serum calcium or albumin-adjusted serum calcium ≥ 2.0 mmol/L (8.0 mg/dL) and ≤ 2.9 mmol/L (11.5 mg/dL)
  * No prior history or current evidence of osteonecrosis of the jaw
  * No Active dental or jaw condition which requires oral surgery, including tooth extraction. Noplanned invasive dental procedures.
* General Laboratory test within normality or with non-relevant deviations of normality as per investigator judgment.
* Patients must have a normal organ and bone marrow function as defined local standards: Leukocytes, Absolute neutrophil count, Platelets, Total bilirubin, AST/ALT/GOT/GPT, Creatinine, Creatinine clearance, Magnesium, Phosphorus.
* Subject with reproductive potential must be willing to use, in combination with her partner, 2 acceptable methods of effective contraception or practice sexual abstinence throughout the study and continue for 6 months after study duration. Subjects who are surgically sterile (e.g. history of bilateral tubal ligation, hysterectomy) or whose sexual partner is sterile (e.g. history of vasectomy) are not required to use additional contraceptive measures".

Exclusion Criteria:

* Invasive breast cancer non-amenable to surgical excision as first therapeutic approach.
* HER2-positive Breast Cancer
* Metastatic breast cancer or other condition that recommends other treatment than surgery as the primary therapeutic approach.
* Prior systemic treatment for any malignancy.
* Treatment with denosumab contraindicated.
* Bleeding diathesis or other concomitant condition that contraindicate inclusion in the study as per investigator judgment.
* High risk of ONJ or hypocalcemia:

  * Inadequate Serum calcium or albumin-adjusted serum calcium < 2.0 mmol/L (8.0 mg/dL) or > 2.9 mmol/L (11.5 mg/dL).
  * Prior history or current evidence of osteonecrosis of the jaw
* Active dental or jaw condition which requires oral surgery, including tooth extraction. Planned invasive dental procedures.
* Subject has known sensitivity to any of the products to be administered during the study (e.g., mammalian derived products, calcium, or vitamin D).
* Subject is pregnant or breast feeding or planning to become pregnant / breastfeed while on study through 6 months after the end of treatment.
* Subject is of child bearing potential and is not willing to use, in combination with her partner, two highly effective methods of contraception or abstinence during treatment and for 5 months after the end oftreatment.
* Patients have prior history or current evidence of osteonecrosis or osteomyelitis of the jaw.
* Patients have active dental or jaw condition which requires oral surgery, including tooth extraction.
* Patients have non-healed dental or oral surgery, including tooth extraction.
* Patients with planned invasive dental procedures for the course of the study.
* Ongoing treatment with denosumab or bisphosphonates

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2022-07-05 (Estimated); Study Completion 2023-02-05 (Estimated)

PRIMARY OUTCOMES:
Antiproliferative and/or pro-apoptotic activity of denosumab | From first biopsy until surgery intervention, which is around four weeks after enrolment
  Changes in the percentage of tumor cells expressing Ki67 and/or cleaved caspase 3 between Biopsy A and Biopsy B.

SECONDARY OUTCOMES:
Correlation between antiproliferative activity of denosumab and Rank/RankL expression | From first biopsy until surgery intervention, which is around four weeks after enrolment
  Modified ratio of Rank/RankL: MR={log(RANK) -1.2} / log(RANKL) as described in Palafox et al [10].
Differential antiproliferative activity of denosumab among the different phenotypes of breast cancers. | From first biopsy until surgery intervention, which is around four weeks after enrolment
  Ki67 estimations for each phenotype
Differential antiproliferative activity of denosumab among pre and post menopausal patients | From first biopsy until surgery intervention, which is around four weeks after enrolment
  Ki67 estimations for each menopausal group
Safety of denosumab and biopsy procedures in terms of Frequency of adverse events (CTCAE V4.) | From first biopsy until surgery intervention, which is around four weeks after enrolment
  Frequency of adverse events derived from denosumab treatment and biopsy procedures

OTHER OUTCOMES:
Changes in overall expression profile determined by RNA expression microarrays | From first biopsy until surgery intervention, which is around four weeks after enrolment
  Changes in rank/rankl normalized expression
Validation of denosumab activity in clinical samples by Trap5b protein expression | From first biopsy until surgery intervention, which is around four weeks after enrolment
  Results compared to preclinical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716